CLINICAL TRIAL: NCT00548171
Title: Evaluation of GSK Biologicals' dTpa Booster Vaccine in Adults, Given 10 Years After Previous dTpa Boosting.
Brief Title: Immunogenicity & Reactogenicity of Boostrix 10 Years After Previous Booster Vaccination in Study NCT01267058
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110804
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Acellular Pertussis; Tetanus; Diphtheria; Diphtheria-Tetanus-acellular Pertussis Vaccines
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — Boostrix

ARMS (2):
- Boostrix I Group (Experimental): Subjects who had received the Boostrix™ vaccine in the primary study 263855/002 (NCT01267058), were boosted in the current study with one dose of the same vaccine, intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Boostrix™
- Boostrix II Group (Active Comparator): Subjects who had received the Td vaccines in the primary study 263855/002 (NCT01267058), were boosted in the current study with one dose of the Boostrix™ vaccine intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Boostrix™

INTERVENTIONS:
Biological: Boostrix™ — Intramuscular injection, 1 dose

SUMMARY:
The purpose of this study is to assess the efficacy and safety of repeating dTpa booster in adults 10 years after previous booster vaccination with dTpa in a previous clinical study (NCT01267058). Only subjects who received the booster vaccination in a previous clinical study are eligible for participation in this study. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

No new recruitment will be performed in this booster phase (see inclusion criteria).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Subjects who have received dTpa vaccine or Td and pa vaccines in study 263855/002 .
* A male or female subject, recruited 10 years (+/- 9 months) after booster vaccination in study 263855/002.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of booster vaccination.
* Written informed consent obtained from the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the booster dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the booster dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to booster vaccination, or planned administration during the active study period
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product
* Previous booster vaccination against diphtheria, tetanus or pertussis since the last dose received in study 263855/002
* History of diphtheria, tetanus, or pertussis diseases.
* Any confirmed or suspected immunosuppressive or immunodeficiency condition, based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the booster dose or planned administration during the study period.
* Occurrence of transient thrombocytopenia or neurological complications following an earlier immunisation against diphtheria and/or tetanus.
* Occurrence of any of the following adverse event after a previous administration of a DTP vaccine :- hypersensitivity reaction to any component of the vaccine; - encephalopathy of unknown aetiology occurring within 7 days following previous vaccination with pertussis-containing vaccine; - fever ≥ 40 °C (axillary temperature) within 48 hours of vaccination not due to another identifiable cause; - collapse or shock-like state within 48 hours of vaccination; - convulsions with or without fever, occurring within 3 days of vaccination.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2007-11-05 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=148

REFERENCES:
- [Background] Booy R, Van der Meeren O, Ng SP, Celzo F, Ramakrishnan G, Jacquet JM. A decennial booster dose of reduced antigen content diphtheria, tetanus, acellular pertussis vaccine (Boostrix) is immunogenic and well tolerated in adults. Vaccine. 2010 Dec 10;29(1):45-50. doi: 10.1016/j.vaccine.2010.10.025. Epub 2010 Oct 23. PMID 20974302
- [Background] Booy R et al. The decennial administration of a reduced antigen content diphtheria, tetanus, acellular pertussis vaccine (dTpa; BoostrixTM) in adults. Abstract presented at IDSA. Philadelphia, USA, 29 October- 1 November 2009.
- [Background] Mertsola J et al. The immunogenicity of repeated administration of reduced-antigen-content dTpa booster in adults. Abstract presented at WSPID. Buenos Aires, Argentina, 19-22 November 2009.
- [Background] Mertsola J et al. The safety of repeated administration of Boostrix™, a reduced-antigen-content dTpa booster. Abstract presented at Excellence In Paediatrics (EIP). Florence, Italy, 3-6 December 2009.
- [Background] Mertsola J et al. The safety of repeated administration of reduced-antigen-content dTpa boosters. Abstract presented at WSPID. Buenos Aires, Argentina, 19-22 November 2009.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110804 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Boostrix I Group | Boostrix II Group
Started | 164 | 39
Completed | 164 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Boostrix I Group | Boostrix II Group | Total
Number analyzed (Participants) | 164 | 39 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.1 (9.98) | 51.0 (8.70) | 50.27 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 33 | 140
  Male | 57 | 6 | 63
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoid (Anti-TT) Antibody Concentrations Equal to or Above (≥) 0.1 International Units Per Milliliter (IU/mL)
Description: Cut-off values defining seroprotected subjects against anti-DT/anti-TT were greater than or equal to (≥) 0.1 IU/mL as assessed by the Enzyme-Linked Immunosorbent Assay (ELISA).
  The analysis was performed and presents results only for subjects who in the previous study NCT01267058, had received the Boostrix™ vaccine as first booster.
Time Frame: One month after the booster vaccination [PI(M1)]
Population: The ATP cohort for immunogenicity included all evaluable subjects who had received the booster dose of Boostrix™ vaccine and for whom immunogenicity data were available. This included subjects for whom assay results were available for antibodies against at least one study vaccine antigen component at the post-vaccination blood-sampling time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 153 | 35
Participants
  Anti-DT ≥ 0.1 PI(M1): number analyzed (Participants) | 152 | 35
  Anti-DT ≥ 0.1 PI(M1) | 151 | 35
  Anti-TT ≥ 0.1 PI(M1) | 153 | 35

2. Secondary Outcome: Number of Subjects With Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations Equal to or Above Cut-off Values
Description: Cut-off values, as assessed by ELISA, were greater than or equal to (≥) 0.1 IU/mL and (≥) 1 IU/mL.
Time Frame: Prior to (PRE) and one month after [PI(M1)] the booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 153 | 35
Participants
  Anti-DT ≥ 0.1 IU/mL, PRE: number analyzed (Participants) | 151 | 34
  Anti-DT ≥ 0.1 IU/mL, PRE | 95 | 20
  Anti-DT ≥ 0.1 IU/mL, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-DT ≥ 0.1 IU/mL, PI(M1) | 151 | 35
  Anti-DT ≥ 1 IU/mL, PRE: number analyzed (Participants) | 151 | 34
  Anti-DT ≥ 1 IU/mL, PRE | 24 | 7
  Anti-DT ≥ 1 IU/mL, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-DT ≥ 1 IU/mL, PI(M1) | 106 | 23
  Anti-TT ≥ 0.1 IU/mL, PRE | 145 | 30
  Anti-TT ≥ 0.1 IU/mL, PI(M1) | 153 | 35
  Anti-TT ≥ 1 IU/mL, PRE | 90 | 23
  Anti-TT ≥ 1 IU/mL, PI(M1) | 153 | 35

3. Secondary Outcome: Anti-diphtheria (Anti-DT) and Anti-tetanus Toxoids (Anti-TT) Antibody Concentrations
Description: Concentrations were presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: Prior to (PRE) and one month after [PI(M1)] the booster vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 153 | 35
IU/mL
  Anti-DT, PRE: number analyzed (Participants) | 151 | 34
  Anti-DT, PRE | 0.200 [0.161 to 0.249] | 0.233 [0.138 to 0.392]
  Anti-DT, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-DT, PI(M1) | 1.889 [1.547 to 2.306] | 1.605 [1.111 to 2.319]
  Anti-TT, PRE | 1.026 [0.859 to 1.224] | 0.845 [0.538 to 1.327]
  Anti-TT, PI(M1) | 6.927 [6.204 to 7.735] | 5.933 [4.768 to 7.384]

4. Secondary Outcome: Number of Subjects With Anti-DT and Anti-TT Antibody Concentrations Equal to or Above Cut-off Values
Description: Cut-off values, as assessed by ELISA, were greater than or equal to (≥) 0.1 IU/mL and ≥ 1 IU/mL.
  This endpoint presents results for subjects included in the ATP cohort for antibody persistence.
Time Frame: Prior (PRE) to booster vaccination
Population: The ATP cohort for antibody persistence included all subjects who had not received any additional dose of DTP vaccine after the booster dose received in study 263855/002 (dTpa-002), with no evidence of diphtheria, tetanus, or pertussis infection or disease, and for whom serological results were available at the pre-booster blood sampling time point
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 160 | 37
Participants
  Anti-DT ≥ 0.1 IU/mL, PRE: number analyzed (Participants) | 158 | 36
  Anti-DT ≥ 0.1 IU/mL, PRE | 102 | 22
  Anti-DT ≥ 1 IU/mL, PRE: number analyzed (Participants) | 158 | 36
  Anti-DT ≥ 1 IU/mL, PRE | 25 | 7
  Anti-TT ≥ 0.1 IU/mL, PRE | 152 | 32
  Anti-TT ≥ 1 IU/mL, PRE | 95 | 25

5. Secondary Outcome: Anti-DT and Anti-TT Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL).
Time Frame: Prior to the booster vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 160 | 37
IU/mL
  Anti-DT, PRE: number analyzed (Participants) | 158 | 36
  Anti-DT, PRE | 0.208 [0.168 to 0.257] | 0.235 [0.144 to 0.384]
  Anti-TT, PRE | 1.031 [0.868 to 1.225] | 0.898 [0.581 to 1.386]

6. Secondary Outcome: Number of Seronegative Subjects for Anti-DT Antibodies - ELISA
Description: Seronegative subjects were defined as subjects with anti-DT antibody concentrations < 0.1 IU/mL prior to vaccination, as assessed by ELISA.
Time Frame: Prior the booster vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 158 | 36
Participants | 56 | 14

7. Secondary Outcome: Number of Seronegative Subjects for Anti-DT Antibodies - Neutralisation Test
Description: Sera with ELISA concentrations <0.1 IU/mL before vaccination were tested for neutralising antibodies using a Vero-cell neutralisation assay. Concentrations ≥0.016 IU/mL by Vero-cell indicated detectable anti-diphteria neutralising antibodies.
Time Frame: Prior the booster vaccination
Population: This analysis was performed on those participants from the According to Protocol (ATP) cohort for antibody persistence who were found to be seronegative for anti-diphtheria antibodies as tested by ELISA.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 56 | 14
Participants | 16 | 4

8. Secondary Outcome: Number of Seropositive Subjects for Anti-pertussis Toxoid (Anti-PT), Anti-filamentous Haemagglutinin (Anti-FHA) and Anti-pertactin (Anti-PRN) Antibodies
Description: Cut-off values, as assessed by ELISA, were greater than or equal to ≥ 5 ELISA Units per millilitre (EL.U/mL) defining seropositive subjects post-vaccination.
Time Frame: Prior the booster vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 160 | 37
Participants
  Anti-PT: number analyzed (Participants) | 160 | 35
  Anti-PT | 137 | 23
  Anti-FHA | 159 | 37
  Anti-PRN: number analyzed (Participants) | 159 | 37
  Anti-PRN | 151 | 33

9. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EL.U/mL)
Time Frame: Prior the booster vaccination
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 160 | 37
EL.U/mL
  Anti-PT: number analyzed (Participants) | 160 | 35
  Anti-PT | 13.9 [11.9 to 16.2] | 8.3 [5.9 to 11.7]
  Anti-FHA | 137.2 [116.7 to 161.3] | 115.6 [80.2 to 166.5]
  Anti-PRN: number analyzed (Participants) | 159 | 37
  Anti-PRN | 56.6 [44.2 to 72.4] | 50.2 [27.9 to 90.4]

10. Secondary Outcome: Number of Seronegative Subjects for Anti-DT Antibodies - ELISA.
Description: as for outcome 6
Time Frame: Prior to the booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 151 | 34
Participants | 56 | 14

11. Secondary Outcome: Number of Seronegative Subjects for Anti-DT Antibodies - Neutralisation Test.
Description: as for outcome 7
Time Frame: Prior to the booster vaccination
Population: This analysis was performed on those participants from the According to Protocol (ATP) cohort for immunogenicity who were found to be seronegative for anti-diphtheria antibodies as assessed by ELISA.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 56 | 14
Participants | 16 | 4

12. Secondary Outcome: Number of Seronegative Subjects for Anti-DT Antibodies - ELISA
Description: as for outcome 6
Time Frame: One month after the booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 152 | 35
Participants | 1 | 0

13. Secondary Outcome: Number of Seronegative Subjects for Anti-DT Antibodies - Neutralisation Test
Description: Sera with ELISA concentrations <0.1 IU/mL before vaccination were tested for neutralising antibodies using a Vero-cell neutralisation assay. Concentrations ≥ 0.016 IU/mL by Vero-cell indicated detectable anti-diphteria neutralising antibodies.
Time Frame: One month after the booster vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 1 | 0
Participants | 0 |

14. Secondary Outcome: Number of Seropositive Subjects for Anti-PT, Anti-FHA and Anti-PRN Antibodies
Description: as for outcome 8
Time Frame: Prior to (PRE) and one month after [PI(M1)] the booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 153 | 35
Participants
  Anti-PT, PRE: number analyzed (Participants) | 153 | 33
  Anti-PT, PRE | 131 | 22
  Anti-PT, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-PT, PI(M1) | 152 | 35
  Anti-FHA, PRE | 152 | 35
  Anti-FHA, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-FHA, PI(M1) | 152 | 35
  Anti-PRN, PRE: number analyzed (Participants) | 152 | 35
  Anti-PRN, PRE | 144 | 31
  Anti-PRN, PI(M1): number analyzed (Participants) | 153 | 34
  Anti-PRN, PI(M1) | 153 | 34

15. Secondary Outcome: Anti-PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EL.U/mL).
Time Frame: Prior to (PRE) and one month after [PI(M1)] the booster vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 153 | 35
EL.U/mL
  Anti-PT, PRE: number analyzed (Participants) | 153 | 33
  Anti-PT, PRE | 13.9 [11.9 to 16.2] | 8.4 [5.9 to 11.8]
  Anti-PT, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-PT, PI(M1) | 126.5 [109.9 to 145.6] | 120.8 [88.9 to 164.2]
  Anti-FHA, PRE | 140.2 [118.9 to 165.4] | 119.3 [81.3 to 175.1]
  Anti-FHA, PI(M1): number analyzed (Participants) | 152 | 35
  Anti-FHA, PI(M1) | 615.3 [543.8 to 696.2] | 677.4 [513.7 to 893.2]
  Anti-PRN, PRE: number analyzed (Participants) | 152 | 35
  Anti-PRN, PRE | 56.2 [43.6 to 72.5] | 45.7 [24.9 to 83.7]
  Anti-PRN, PI(M1): number analyzed (Participants) | 153 | 34
  Anti-PRN, PI(M1) | 303.6 [259.6 to 355.0] | 370.7 [280.5 to 489.9]

16. Secondary Outcome: Number of Subjects With Booster Response to Anti-PT, Anti-FHA and Anti-PRN
Description: Booster response was defined as appearance of antibodies in subjects who were seronegative at the pre-vaccination time point (i.e. with concentrations < 5 El.U/mL) or at least 2-fold increase of pre-vaccination antibody concentrations in subjects who were seropositive at the pre-vaccination time point (i.e. with concentrations ≥5 El.U/mL).
Time Frame: One month after the booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix I Group | Boostrix II Group
Number analyzed (Participants) | 152 | 35
Participants
  Anti-PT: number analyzed (Participants) | 152 | 33
  Anti-PT | 148 | 33
  Anti-FHA | 119 | 31
  Anti-PRN: number analyzed (Participants) | 152 | 34
  Anti-PRN | 106 | 26

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Relationship analysis was not performed.
  For safety assessment Boostrix I Group and Boostrix II Group were pooled into Booster Pooled Group.
Time Frame: During the 4-day (Day 0-3) follow-up period after booster vaccination
Population: The Total Vaccinated Cohort (TVC) included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Groups:
- Boostrix Pooled Group: Subjects who had received the Boostrix™ and the Td vaccines in the primary study 263855/002 (NCT01267058) administrated intramuscularly in the deltoid region of the non-dominant arm were boosted in the current study with one dose of Boostrix™ vaccine, intramuscularly in the deltoid region of the non-dominant arm.
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 203
Participants
  Any Pain | 142
  Grade 3 Pain | 2
  Any Redness | 72
  Grade 3 Redness | 14
  Any Swelling | 66
  Grade 3 Swelling | 20

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache, gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
  For safety assessment Boostrix I Group and Boostrix II Group were pooled into Booster Pooled Group.
Time Frame: During the 4-day (Day 0-3) follow-up period after booster vaccination
Population: The Total Vaccinated Cohort (TVC) included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 203
Participants
  Any Fatigue | 47
  Grade 3 Fatigue | 0
  Related Fatigue | 25
  Any Fever | 6
  Grade 3 Fever | 0
  Related Fever | 5
  Any Gastrointestinal symptom | 15
  Grade 3 Gastrointestinal symptom | 1
  Related Gastrointestinal symptom | 7
  Any Headache | 39
  Grade 3 Headache | 2
  Related Headache | 18

19. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
  For safety assessment Boostrix I Group and Boostrix II Group were pooled into Booster Pooled Group.
Time Frame: During the 31-day (Day 0-30) follow-up period after booster vaccination
Population: The Total Vaccinated Cohort (TVC) included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 203
Participants | 35

20. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
  For safety assessment Boostrix I Group and Boostrix II Group were pooled into Booster Pooled Group.
Time Frame: Following the booster vaccination
Population: The Total Vaccinated Cohort (TVC) included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Pooled Group
Number analyzed (Participants) | 203
Participants | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4-day (Days 0-3) follow-up period post booster vaccination; Unsolicited AEs: during the 31-day (Days 0-30) follow-up period post booster vaccination; SAEs: during the entire study period (following booster vaccination).
Description: For safety assessment Boostrix I Group and Boostrix II Group were pooled into Booster Pooled Group.
Arm/Group | Boostrix Pooled Group
All-Cause Mortality (participants affected / at risk) | 0/203
Serious Adverse Events (participants affected / at risk) | 0/203
Other Adverse Events (participants affected / at risk) | 163/203
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Pooled Group (N=203)
Fatigue (General disorders) | 47 (47)
Gastrointestinal disorder (Gastrointestinal disorders) | 15 (15)
Headache (Nervous system disorders) | 40 (40)
Pain (General disorders) | 142 (142)
Erythema (Skin and subcutaneous tissue disorders) | 72 (72)
Swelling (General disorders) | 66 (66)
Injection site pruritus (General disorders) | 9 (9)
Pyrexia (General disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.